CLINICAL TRIAL: NCT03291548
Title: Effect of a Quinoa-enriched Biscuit as Novel Food Product to Improve CVD Risk Markers in Older Adults: a Randomised Crossover Study
Brief Title: Quinoa Biscuit & CVD Risk Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: The Regional Centre for Studies in Food and Health (CREAS), Valparaíso, Chile (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UREC/16/0106
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Diseases; Dyslipidemias; Lipid Profile
Keywords: Quinoa; Functional food; Cardiovascular disease; Cholesterol; Lipid profile; Randomised Control Trial
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind: researcher and particiapant unaware of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quinoa Biscuit (Experimental): The quinoa-enriched biscuits containing 7.11g quinoa flour.
  Interventions: Dietary Supplement: Quinoa biscuit
- Control biscuit (Placebo Comparator): The placebo control biscuit: an iso-energetic, matched product in terms of appearance, taste, texture and smell.
  Interventions: Dietary Supplement: Control biscuit

INTERVENTIONS:
Dietary Supplement: Quinoa biscuit — 2x15g biscuits per day for 28 consecutive days (4 weeks).
  Arms: Quinoa Biscuit
Dietary Supplement: Control biscuit — 2x15g biscuits per day for 28 consecutive days (4 weeks).
  Arms: Control biscuit

SUMMARY:
Cardiovascular disease (CVD) is one of the most common chronic diseases in older populations, which has been increasing in line with rising overweight and obesity levels in recent years. Dietary intake is a major modifiable risk factor for CVD, and one such recommendation is to increase the intake of essential (omega-3) polyunsaturated fats in our diets, for example by consuming more oily fish. We know, however, from large population level dietary surveys, that many individuals within the United Kingdom (UK) population are not consuming enough oily fish. Therefore, alternative dietary sources of omega-3 polyunsaturated fats are required to help meet consumer needs.

Quinoa is a traditional Andean seed crop consumed in a similar fashion to staple cereal grains in Europe, and the popularity of quinoa has been growing worldwide because of its nutritional content and perceived healthiness. Quinoa contains a small amount of fat, but the ratio of omega-6 and omega-3 essential fats is more favourable in quinoa than in other plant oils. An opportunity therefore exists to incorporate quinoa flour into more frequently consumed food products (e.g. biscuits) as an alternative means of increasing consumers omega-3 intake.

The purpose of this study is to investigate the effect of consuming quinoa-enriched biscuits, compared to control, on markers of CVD risk over 4-weeks in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Free-living, apparently healthy adults
* Aged 50-75 years at recruitment
* Low fish consumers (<2 servings/wk)
* Non-smokers
* Not regularly consuming plant stanols

Exclusion Criteria:

* Non-free-living adults
* Aged <50 or >75 years at recruitment
* Fish consumers (2 servings/wk or more)
* Current smokers
* Pregnant/lactating females
* Coeliac disease, wheat intolerance or any other food allergy or intolerance that would prevent consumption of the biscuits
* Currently taking any fish oil-containing supplement
* Diagnosed with a chronic medical condition (such as diabetes; CVD autoimmune/ inflammatory disorders; cancer)
* Prescribed cholesterol or blood pressure lowering medications
* Daily consumption of plant stanols

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | Change from baseline compared to control arm
  Plasma cholesterol

SECONDARY OUTCOMES:
Triglycerides | Change from baseline compared to control arm
  measured in plasma
LDL-cholesterol | Change from baseline compared to control arm
  measured in plasma
HDL-cholesterol | Change from baseline compared to control arm
  measured in plasma
total/HDL-cholesterol ratio | Change from baseline compared to control arm
  measured in plasma
Poly-unsaturated fatty acid status | Change from baseline compared to control arm
  measured in plasma
Antioxidant status | Change from baseline compared to control arm
  Ferric-reducing Ability Plasma
Inflammatory status | Change from baseline compared to control arm
  C-reactive protein
Blood pressure | Change from baseline compared to control arm
  Diastolic and systolic
Weight | Change from baseline compared to control arm
  Kg

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pourshahidi LK, Caballero E, Osses A, Hyland BW, Ternan NG, Gill CIR. Modest improvement in CVD risk markers in older adults following quinoa (Chenopodium quinoa Willd.) consumption: a randomized-controlled crossover study with a novel food product. Eur J Nutr. 2020 Oct;59(7):3313-3323. doi: 10.1007/s00394-019-02169-0. Epub 2020 Jan 9. PMID 31919583